CLINICAL TRIAL: NCT00370669
Title: Effect of Intravitreal Bevacizumab on Clinically Significant Macular Edema
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8411
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2007-02

CONDITIONS: Diabetic Macular Edema
Keywords: Bevacizumab; CSME; MPC; Triamcinolone acetonide
MeSH Terms: interventions — Bevacizumab; Triamcinolone Acetonide

INTERVENTIONS:
Drug: bevacizumab
Drug: triamcinolone acetonide

SUMMARY:
to compare the effect of intravitreal bevacizumab alone or in combination with triamcinolone acetonide with laser photocoagulation on clinically significant macular edema (CSME)

DETAILED DESCRIPTION:
we entered 150 eyes into the study that recruitment of cases finished recently.Eligible eyes randomly assign to one of the study arms including intravitreal bevacizumzb, intravitreal bevacizumzb/triamcinolone and macular photocoagulation groups. Every patient needs at least 1 year followup. During this time BCVA, OCT, FA will be done for each patient and inaccording to interpretation of datas and fundus exam repeatation of injection will be done.

ELIGIBILITY:
Inclusion Criteria:

* case with clear media IOP below 23 mm/Hg female after menopause at least for 12 months or had 2 contraceptive roots visual acuity between 20/50 to 20/320

Exclusion Criteria:

* no PRP or N.d YAG laser in past 6 months no intraocular surgery in past 12 months
* CVA in past 12 months blood sugar above 250
* active infection in extraocular adnexa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2005-11; Study Completion 2007-02

PRIMARY OUTCOMES:
visual acuity
central macular thickness

SECONDARY OUTCOMES:
Leakage in fluorescein angiography
intraocular pressure
cataract progression
anterior chamber reaction

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soheilian, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Masoud Soheilian, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Soheilian M, Garfami KH, Ramezani A, Yaseri M, Peyman GA. Two-year results of a randomized trial of intravitreal bevacizumab alone or combined with triamcinolone versus laser in diabetic macular edema. Retina. 2012 Feb;32(2):314-21. doi: 10.1097/IAE.0b013e31822f55de. PMID 22234244
- [Derived] Soheilian M, Ramezani A, Obudi A, Bijanzadeh B, Salehipour M, Yaseri M, Ahmadieh H, Dehghan MH, Azarmina M, Moradian S, Peyman GA. Randomized trial of intravitreal bevacizumab alone or combined with triamcinolone versus macular photocoagulation in diabetic macular edema. Ophthalmology. 2009 Jun;116(6):1142-50. doi: 10.1016/j.ophtha.2009.01.011. Epub 2009 Apr 19. PMID 19376585